CLINICAL TRIAL: NCT05474781
Title: Micro-elimination of HCV Infection Among People Who Use Drug (PWUD) in British.Columbia: A Comprehensive, Multidisciplinary, Scalable Programmatic Approach
Brief Title: Eliminating HCV Infection Among PWUD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vancouver Infectious Diseases Centre (Other)
Responsible Party: Sponsor
Other Study IDs: IN-CA-987-5437
Record Dates: First submitted 2022-07-07; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis C, Chronic; Drug Use
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Epclusa — HCV treatment

SUMMARY:
Identify 300 PWUD with chronic, viremic HCV infection and engage them in a multidisciplinary, generalizable model of care and initiate HCV treatment

ELIGIBILITY:
Inclusion Criteria:

1. Ability to review, sign and date the IRB/IEC approved informed consent form
2. Age ≥19 years
3. Documented HCV RNA positive for 6 months or more, with any HCV genotype
4. Active PWUD (ongoing drug use or documented use within the previous 6 months) OR active enrolment in an opiate substitution program

Exclusion Criteria:

1. Previous DAA-based HCV treatment
2. Pregnant or breast-feeding
3. Indications of decompensated liver disease
4. Diagnosis of active hepatocellular carcinoma
5. Positive test at the time of screening for hepatitis B surface antigen (HBsAg)
6. Frequent injecting drug use that is judged by the treating physician to compromise subsequent HCV treatment safety
7. Inability or unwillingness to provide informed consent or to actively engage in care leading to the initiation of HCV treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV-infected current drug users
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of individuals enrolled in the study who initiate HCV treatment | 60 months

SECONDARY OUTCOMES:
The proportion of individuals enrolled in the study who achieve sustained virologic response | 72 months

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver Infectious Diseases Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No